CLINICAL TRIAL: NCT03632694
Title: Replacing Sedentary Time With Light Activity
Brief Title: The Move for Your Health Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cindy Blair, PhD, MPH (Other)
Collaborators: University of New Mexico Cancer Center (Other); American Cancer Society, Inc. (Other)
Responsible Party: Sponsor-Investigator, Cindy Blair, PhD, MPH, Principal Investigator, University of New Mexico
Organization: University of New Mexico (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 16-003; INST UNM 1520 (Other: UNM)
Record Dates: First submitted 2018-08-08; First posted 2018-08-15 (Actual); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Cancer
Keywords: cancer survivor; cancer survivorship; light physical activity; sedentary behavior; mHealth; Jawbone
MeSH Terms: conditions — Neoplasms; Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: 3-arm randomized controlled trial; participants were block randomized with equal allocation to 3 arms within 2 strata defined by body mass index (BMI; <30 vs. >=30 kg/m2)
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Health Coaching and Tech Support (Experimental): Participants receive tech support for using the "Jawbone UP2" activity monitor and smartphone app, and education materials and health coaching to achieve their goals to reduce sedentary time and increase their daily steps.
  Interventions: Behavioral: Health Coaching and Tech Support
- Tech Support Only (Active Comparator): Participants receive tech support for using the "Jawbone UP2" activity monitor and smartphone app and education materials on reducing sedentary behavior.
  Interventions: Behavioral: Tech Support Only
- Waitlist Control (No Intervention): Participants are instructed to maintain their regular activities. Upon completion of the 16-week intervention, participants receive the "Jawbone UP2" activity monitor, education materials, and one session of tech support/health coaching.

INTERVENTIONS:
Behavioral: Health Coaching and Tech Support — Participants will receive a "Jawbone UP2" activity monitor and education materials about the negative consequences of sedentary behavior and suggestions for breaking up sedentary time with light physical activity. Participants receive 5 telephone coaching calls to set up the "Jawbone UP2" monitor with their smartphone app and receive tech support help with changing the settings/goals on the app. Additionally, this arm receives health coaching to provide encouragement and further motivate and help study participants to modify their sedentary behavior.
  Arms: Health Coaching and Tech Support
Behavioral: Tech Support Only — Participants will receive a "Jawbone UP2" activity monitor and education materials about the negative consequences of sedentary behavior and suggestions for breaking up sedentary time with light physical activity. Participants receive 5 telephone coaching calls to set up the "Jawbone UP2" monitor with their smartphone app and receive tech support help with changing the settings/goals on the app. However, there is no additional health coaching.
  Arms: Tech Support Only

SUMMARY:
The Move for Your Health Pilot Study is a 16-week study in older cancer survivors to replace and break-up sedentary activity with short bouts of light physical activity.

DETAILED DESCRIPTION:
This pilot study will determine the feasibility and acceptability of a mobile health (mHealth) intervention to replace and break-up sedentary time with intermittent bouts of light physical activity. The intervention uses an electronic activity monitor ("Jawbone UP2"; worn on the wrist) that pairs with a mobile app, which together promote awareness and enable self-monitoring of both physical activity (steps per day) and inactivity (wristband gently vibrates after a specified time of inactivity). Pre-post intervention change in objective, subjective, and biologic data will be compared between groups.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 years or older at the time of enrollment
* Diagnosed with local or regionally staged cancer (any site) and completed primary treatment
* Own a smartphone capable of running the "Jawbone UP2" app
* Willingness to be randomized to any of the 3 study arms, attend 2 clinic visits, and wear activity monitors (activPAL and actiGraph) at weeks 1 and 16 for 7 days; "Jawbone UP2" wristband monitor during weeks 2-16 during waking hours.
* Able to read, speak, and understand English.
* Living independently and capable of walking 3 blocks (approximately 1300 steps or 0.25 mile) without an assistive device (e.g., cane, walker)
* Residence within Bernalillo County or the four surrounding counties (to reduce travel burden)

Exclusion Criteria:

* Currently participating in a program to decrease sedentary time or increase physical activity
* Paid employment or volunteer position for greater than 20 hours per week
* Severe impairments or pre-existing medical limitations for engaging in daily light physical activity
* Wrist size >20 cm

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2016-07-06 (Actual); Primary Completion 2017-07-20 (Actual); Study Completion 2017-07-20 (Actual)

PRIMARY OUTCOMES:
Change in total volume of sedentary time (hours/day) | Baseline to 16-weeks
  Change in the average number of hours/day of sedentary time measured over a 1-week period using activPAL, at both baseline and 16-weeks post-intervention
Change in the number of breaks in sedentary time | Baseline to 16-weeks
  Change in the average number of breaks in sedentary time measured over a 1-week period using activPAL, at both baseline and 16-weeks post-intervention

SECONDARY OUTCOMES:
Change in light physical activity | Baseline to 16-weeks
  Change in the average number of hours per day spent in light physical activity (or higher intensity) measured over a 1-week period using activPAL, at both baseline and 16-weeks post-intervention
Change in steps per day | Baseline to 16-weeks
  Change in the average number of steps per day measured over a 1-week period using activPAL, at both baseline and 16-weeks post-intervention
Change in physical performance | Baseline to 16-weeks
  Change in the average physical performance score as measured by the Short Physical Performance Battery (SPPB). This performance battery includes chair stands, balance tests, and the 8-foot usual gait speed. Each subscale score ranges from 0 (cannot do) to 4 (good performance). The subscales are summed for a total score, which ranges from 0 (lowest level of performance) to 12 (highest level of performance)
Change in physical functioning (ranging from basic to strenuous activities) | Baseline to 16-weeks
  Change in self-reported physical functioning as measured by the 36-item Short Form Survey (SF-36) physical functioning subscale. Raw scores range from 0 (worst functioning) to 100 (best functioning)
Change in health-related quality of life (self-reported mental, physical, and social health and well-being) | Baseline to 16-weeks
  Change in quality of life as measured by the SF-36; each of the 8 subscales and 2 component summary scores; scores based on proprietary algorithm from Optum; higher scores represent better quality of life)
Change in cardiometabolic markers | Baseline to 16-weeks
  Change in fasting glucose, insulin and lipids, as well as high-sensitivity C-Reactive Protein (CRP)

CONTACTS AND LOCATIONS:
Overall Officials: Cindy K Blair, PhD, MPH, Principal Investigator — University of New Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Blair CK, Harding E, Wiggins C, Kang H, Schwartz M, Tarnower A, Du R, Kinney AY. A Home-Based Mobile Health Intervention to Replace Sedentary Time With Light Physical Activity in Older Cancer Survivors: Randomized Controlled Pilot Trial. JMIR Cancer. 2021 Apr 13;7(2):e18819. doi: 10.2196/18819. PMID 33847588